CLINICAL TRIAL: NCT03247569
Title: Non-interventional Study on Edoxaban Treatment in Routine Clinical Practice for Patients With Non-valvular Atrial Fibrillation (ETNA-AF-Thailand)
Brief Title: Edoxaban Treatment in Routine Clinical Practice for Patients With Non-Valvular Atrial Fibrillation (NVAF)
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Thailand) Ltd., a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DU176b-C-A4011
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular Atrial Fibrillation; Real World Evidence; Observational Safety
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Edoxaban: Patients treated with Edoxaban
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Edoxaban according to Package Information (Summary of Product Characteristics (SmPC)).
  Other Names: Lixiana

SUMMARY:
In order to understand the risks and benefits of edoxaban use in a real-world clinical setting in the NVAF indication, Daiichi-Sankyo Thailand proposed this non-interventional study (NIS) to gain insight into the safety (bleeding, liver adverse events, all-cause mortality and other adverse events) of edoxaban use in non-preselected patients with NVAF.

DETAILED DESCRIPTION:
Edoxaban was recently approved by The Thai Food and Drug Administration (Thai FDA) (date: 2nd December 2016) for the prevention of stroke and systemic embolism in adult patients with NVAF with one or more risk factors, such as congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, prior stroke or transient ischemic attack (TIA). Treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) and prevention of recurrent DVT and PE in adults.

In order to understand the risks and benefits of edoxaban use in a real-world clinical setting in the NVAF indication, Daiichi-Sankyo Thailand proposed this non-interventional study (NIS) to gain insight into the safety (bleeding, liver adverse events, all-cause mortality and other adverse events) of edoxaban use in non-preselected patients with NVAF.

Real world evidence data of routine clinical practice use of edoxaban up to 2 years will be collected and evaluated in approximately 300 patients, treated by specialized as well as non-specialized physicians in hospital centres.

ELIGIBILITY:
Inclusion Criteria:

* Is a NVAF-patient whose physician has made the clinical decision to prescribe edoxaban therapy according to Package Information
* Has provided written informed consent to participate in the study

Exclusion Criteria:

* Is participating in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary strategy is to include only patients with NVAF who are to be treated with edoxaban according to Package Information (Summary of Product Characteristics (SmPC)). To ensure that the physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban.
  Patients must have provided written informed consent for participation in the study (ICF) and should not participate simultaneously in any interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with real world safety events | 2 years

SECONDARY OUTCOMES:
Number of participants with patient relevant outcomes | 2 years
  Categories: Strokes (ischaemic and haemorrhagic), Systemic Embolic Events (SEE), Transient Ischemic Attack (TIA), Major Adverse Cardiovascular Events (MACE), Venous Thromboembolism (VTE), Acute Coronary Syndrome (ACS), Hospitalisations related to cardiovascular (CV) condition
Average duration of exposure to edoxaban | within 2 years
Number of participants compliant with edoxaban therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Late Phase Operations Lead, Global Medical Affairs, Study Director — Daiichi Sankyo (Thailand) Ltd., a Daiichi Sankyo Company; Study Project Manager, Study Chair — Daiichi Sankyo (Thailand) Ltd., a Daiichi Sankyo Company
Locations (6):
- Thailand (6):
  - Srinagarind Hospital and Queen Sirikit Heart Center of the Northeast, Khon Kaen, Muang District
  - Bangkok Heart Hospital, Bangkok
  - Bhumibol Adulyadej Hospital, Bangkok
  - Bangkok Hospital Chiang Mai, Chiang Mai
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Thammasat University Hospital, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Derived] De Caterina R, Unverdorben M, Chen C, Choi EK, Koretsune Y, Morrone D, Pecen L, Bramlage P, Wang CC, Yamashita T, Kirchhof P. Two-Year Follow-Up of Patients With Atrial Fibrillation Receiving Edoxaban in Routine Clinical Practice: Results From the Global ETNA-AF Program. Clin Cardiol. 2025 Feb;48(3):e70091. doi: 10.1002/clc.70091. PMID 40014354